CLINICAL TRIAL: NCT01008111
Title: The Effect of a Sodium Bicarbonate and Hydrogen Peroxide Gel on Wound Healing of Incisional Wounds for Bilateral Hernia Repair
Brief Title: Wound Healing of Incisional Wounds for Bilateral Hernia Repair
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study never initiated
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00009521
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-01

CONDITIONS: Wound Healing
Keywords: regeneration; tissue survival; biological processes; connective tissue; tissue
MeSH Terms: interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrogen Peroxide Oxygen producing gel (Active Comparator): On Day 0 patients will undergo bilateral inguinal surgery. One side will be dressed using a standard surgical dressing, while the other will use a combination hydrogen peroxide/baking soda gel placed over the wound and covered with a sealing dressing. The study team will determine which side gets assigned standard surgical dressing by the flip of a coin.
  Interventions: Drug: Hydrogen Peroxide Oxygen producing gel
- Dermabond-Placebo Comparator (Placebo Comparator): On Day 0 patients will undergo bilateral inguinal surgery. One side will be dressed using a standard surgical dressing, while the other will use a combination hydrogen peroxide/baking soda gel placed over the wound and covered with a sealing dressing. The study team will determine which side gets assigned standard surgical dressing by the flip of a coin.
  Interventions: Drug: Dermabond

INTERVENTIONS:
Drug: Dermabond — On Day 0 patients will undergo bilateral inguinal surgery. One side will be dressed using a standard surgical dressing, while the other will use a combination hydrogen peroxide/baking soda gel placed over the wound and covered with a sealing dressing. The study team will determine which side gets assigned standard surgical dressing by the flip of a coin.
  Arms: Dermabond-Placebo Comparator
Drug: Hydrogen Peroxide Oxygen producing gel — On Day 0 patients will undergo bilateral inguinal surgery. One side will be dressed using a standard surgical dressing, while the other will use a combination hydrogen peroxide/baking soda gel placed over the wound and covered with a sealing dressing. The study team will determine which side gets assigned standard surgical dressing by the flip of a coin.
  Arms: Hydrogen Peroxide Oxygen producing gel

SUMMARY:
The purpose of this research study is to test the safety of an oxygen producing gel (produced by combining baking soda and hydrogen peroxide) and see what effects (good and bad) it has on skin incisions in children.

Baking soda and hydrogen peroxide have been approved by the US Food and Drug Administration (FDA), but have not been approved for use in this manner.

It is hypothesized that a combination of sodium bicarbonate and hydrogen peroxide may enhance wound healing of incisional wounds for bilateral hernia repair.

DETAILED DESCRIPTION:
Wound healing is a complex regeneration process, which is characterized by degradation and re-assembly of connective tissue and epidermal layer. The pH value within the wound-milieu influences indirectly and directly all biochemical reactions taking place in this process of healing. Interestingly, it is so far a neglected parameter for the overall outcome. For more than three decades the common assumption amongst physicians was that a low pH value, such as it is found on normal skin, is favorable for wound healing. However, investigations have shown that in fact some healing processes such as the take-rate of skin-grafts require an alkaline milieu. The matter is thus much more complicated than it was assumed.

One review drew the conclusion that wound pH is potent influential factor for the healing process and that different pH ranges are required for certain distinct phases of wound healing. Further systematic data needs to be collected for a better understanding of the pH requirements under specific circumstances. This is important as it will help to develop new pH targeted therapeutic strategies. Such shifts in the pH can be accomplished through the use of sodium biocarbonate (baking soda)

Another common agent used in wound treatments is hydrogen peroxide. It has been hypothesized that hydrogen peroxide would accelerate reepithelization and/or have a positive effect on infection. However, the results of using hydrogen peroxide alone do not appear to support this hypothesis. (Table 1)

However, one report using a combination of baking soda and hydrogen peroxide on post-surgical wound healing showed a significant increase in wound healing from oral surgery. A randomized, double-blind crossover study involving 25 patients requiring bilateral maxillary gingival flap surgery was completed. The effects of twice daily brushing with a baking soda-hydrogen peroxide dentifrice or a placebo dentifrice were observed over a 28-day post-surgical period. At days 7 and 14, soft tissue appearance/wound healing (STA) was assessed based on color and edema,. Post-surgical wound healing was statistically significantly improved at day 7 with the trend continuing to day 14 when sodium bicarbonate-hydrogen peroxide was used as compared to a control. Such materials were shown to be a possibly effective aid in the early phase of healing following gingival flap surgery. It has been determined that this combination of products may increase oxygen content to the wound sites.

ELIGIBILITY:
Inclusion Criteria:

* Children with surgery requiring bilateral similar inguinal incisions (i.e. bilateral orchidopexy, bilateral hernia repair).

Exclusion Criteria:

None.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Wound infection, wound dehiscence, allergic reaction to gel components, width, elevation, color, marks and general appearance measured at clinic visits. | days7 and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hodges, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided